CLINICAL TRIAL: NCT03401749
Title: Efficacy of Preadmission Theraworx Wipe Use for Surgical Site Infection Prophylaxis in Adult Orthopaedic Surgery Patients: A Randomized Controlled Trial
Brief Title: Preadmission Skin Wipe Use for Surgical Site Infection Prophylaxis in Adult Orthopaedic Surgery Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding issues, poor recruiting and compliance of the patients.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ashish Shah, Assistant Professor, Department of Orthopaedics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-300000508
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control Group (No Intervention): Usual preadmission surgery instructions (shower the night before).
- Theraworx Group (Experimental): Usual preadmission surgery instructions (shower the night before) plus theraworx skin wipe system use the night before surgery and 1 hour before surgery.
  Interventions: Other: Theraworx Bath Wipes
- CHG Group (Experimental): Usual preadmission surgery instructions (shower the night before) plus chlorhexidine gluconate (CHG) skin wipe system use the night before surgery and 1 hour before surgery.
  Interventions: Drug: Chlorhexidine Gluconate 2% Wipe

INTERVENTIONS:
Drug: Chlorhexidine Gluconate 2% Wipe — Patients will be instructed to use CHG wipes after showering the night before surgery and again on the morning of surgery.
  Arms: CHG Group
Other: Theraworx Bath Wipes — Theraworx TM is a cosmetic product that is a non-rinse skin formulation that combines multiple ingredients, including Aloe Concentrate, Allantoin, Tego Betaine F 50, Tego Betaine L-7, Lauryl Glucoside, Abil 8852, Vitamin E, Natural Fragrances, Methyl paraben, Propyl paraben, EDTA, Antimicrobial Preservative, Colloidal Silver, and Beta Glucan, in preoperative disposable bath wipes. The main proposed antimicrobial mechanism of action involves the local reduction in skin pH to around 4.6.
  Other Names: Theraworx
  Arms: Theraworx Group

SUMMARY:
Intervention: This study will involve three different study arms with different interventions prior to surgery: (1) shower only, (2) shower plus Theraworx wipes, (3) shower plus chlorhexidine wipes

Study Design: Single center RCT

Sample Size: 500 patients, aged 18+

Objectives: Primary Objectives:

1. Monitor for safety and adverse effects.
2. Evaluate for differences in peri-operative skin cultures between treatment groups;
3. Compare surgical site infection rates between groups.

Secondary Objectives:

1. Assess for patient compliance for each different treatment arms.
2. Measure patient satisfaction.
3. Measure nurse satisfaction.
4. Visual assessment of wound healing

Expected Results: We expect no statistically significant difference in peri-operative cultures or surgical site infection rates between groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient between ages 18-64
* Scheduled and deemed healthy enough to undergo orthopaedic surgery
* Willing and able to comply with protocol

Exclusion Criteria:

* Clinical signs of infection
* Contraindication to CHG or Theraworx
* Previous allergic reaction to CHG or Theraworx
* Surgeon's Discretion

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ashish shah, md, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Highlands Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Theraworx Group | CHG Group
Started | 59 | 67 | 77
Completed (Completion was determined as patients who completed the 2 week, 6 week, and 3 month postoperative surgical site questionnaire. If patients did not complete all 3 post operative questionnaires, they were marked as "lost to follow up". This does not suggest any adverse event occurred, simply that patients stopped coming to their postoperative clinical visits.) | 39 | 51 | 51
Not Completed | 20 | 16 | 26
Not completed — Lost to Follow-up | 20 | 16 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Theraworx Group | CHG Group | Total
Number analyzed (Participants) | 59 | 67 | 77 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 59 | 59 | 160
  >=65 years | 17 | 8 | 18 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (14.92) | 49.71 (14.93) | 49.68 (14.95) | 51.66 (14.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 44 | 52 | 136
  Male | 19 | 23 | 25 | 67
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 59 | 67 | 77 | 203
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Average BMI of each cohort.
  kg/m^2 | 32.46 (7.58) | 33.61 (7.92) | 32.8 (7.59) | 33.15 (7.86)
Tobacco Use [Count of Participants; unit: Participants] — Participants that recorded previous or current use of tobacco products.
  Participants | 19 | 24 | 28 | 71
Presence of Diabetes [Count of Participants; unit: Participants] — Number of participants with a diagnosis of diabetes.
  Participants | 10 | 14 | 14 | 38
Hypertension [Count of Participants; unit: Participants] | 38 | 37 | 43 | 118
Presence of Rheumatoid Arthritis [Count of Participants; unit: Participants] — Number of participants with a diagnosis of Rheumatoid Arthritis
  Participants | 6 | 0 | 8 | 14
Presence of Preoperative Neuropathy [Count of Participants; unit: Participants] — Number of participants who have a diagnosis of neuropathy affecting the lower limb.
  Participants | 7 | 7 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Developed a Surgical Site Infection
Description: Clinical development of a surgical site infection in the postoperative period.
Time Frame: Within 1 year of Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Theraworx Group | CHG Group
Number analyzed (Participants) | 59 | 67 | 77
Participants | 2 | 1 | 3

2. Secondary Outcome: Number of Patients Compliant With the Requirement of Their Study Group
Description: Survey on patient's ability to follow the study guidelines. For example, if the patient was placed in the Theraworx study group, did they properly follow the instructions to shower and use the Theraworx skin wipe system the night before surgery.
Time Frame: Day before and day of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Theraworx Group | CHG Group
Number analyzed (Participants) | 59 | 67 | 77
Participants | 45 | 66 | 67

ADVERSE EVENTS:
Time Frame: Adverse events (i.e surgical site infection) were recorded if they occurred within one year from the date of surgery.
Description: Upon completion of this study, we retrospectively observed the occurrence of any adverse event in our patient population utilizing our electronic medical record. . Using the standardized clinical trials definition of "adverse event" we carefully determined the rate at which these events occurred.
Arm/Group | Control Group | Theraworx Group | CHG Group
All-Cause Mortality (participants affected / at risk) | 2/59 | 1/67 | 1/77
Serious Adverse Events (participants affected / at risk) | 2/59 | 1/67 | 1/77
Other Adverse Events (participants affected / at risk) | 2/59 | 1/67 | 3/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=59) | Theraworx Group (N=67) | CHG Group (N=77)
Exacerbated Congestive Heart Failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) — Patient with history of CHF suffered from acute exacerbation in within the 1 year postoperative time frame.
Carotid Pseudo-aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Number of patients who suffered from a carotid pseudo-aneurysm in the 1 year postoperative time frame.
Pulmonary Embolism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Number of patients who developed a pulmonary embolism within 1 year from their date of surgery.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=59) | Theraworx Group (N=67) | CHG Group (N=77)
Surgical Site Infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) — This is the same measure as the primary outcome "number of participants who developed a surgical site infection"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT03401749/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT03401749/SAP_001.pdf
  • Informed Consent Form (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT03401749/ICF_002.pdf